CLINICAL TRIAL: NCT07369609
Title: Investigation of Factors Affecting Physical Activity Level in Children With Duchenne Muscular Dystrophy Based on the International Classification of Functioning, Disability and Health - Child and Youth Version
Brief Title: Factors Influencing Physical Activity Levels in Children With Duchenne Muscular Dystrophy: An ICF-CY-Based Study
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Serenay Zorlu, Research Assistant, Ankara Medipol University
Other Study IDs: FTREK25/64
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: duchenne muscular dystrophy; physical activity; ICF-CY
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is a neuromuscular disease characterized not only by progressive muscle weakness but also by cognitive, behavioral, and psychosocial impairments. Motor losses that occur during disease progression reduce physical activity levels in children and increase the risk of developing a sedentary lifestyle. Interventions aimed at maintaining or promoting physical activity in children with DMD are important for preventing secondary complications associated with disuse and physical inactivity. To develop effective interventions, there is a need for comprehensive knowledge regarding the factors that influence physical activity levels.

Current literature indicates that, in typically developing children, physical activity levels are influenced not only by motor factors but also by cognitive status, sleep, behavioral characteristics, and family-related environmental and psychosocial factors. However, information regarding these multidimensional factors affecting physical activity levels in children with DMD remains limited.

This study aims to identify the body functions, activity, participation, environmental, and personal factors affecting physical activity levels in children with DMD based on the framework of the International Classification of Functioning, Disability and Health - Children and Youth Version (ICF-CY). Accordingly, the effects of posture, functional capacity, ambulatory status, balance, other musculoskeletal parameters, cognitive status, sleep habits and sleep quality, fear of falling, and behavioral characteristics, as well as family-related factors including parenting style, perceptions of physical activity, stress level, attitudes and perceptions toward daily life events, and disease impact, will be evaluated. The impact of these variables on physical activity levels and the magnitude of this effect will be examined within the ICF-CY framework.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common inherited neuromuscular disorder, affecting approximately one in 3,500-5,000 live male births worldwide. It is caused by various mutations in the dystrophin gene located on Xp21.2, most commonly deletions and duplications, leading to the absence of dystrophin protein in skeletal muscle, cardiac muscle, and the central nervous system. The lack of dystrophin results in progressive muscle weakness beginning in early childhood, typically between 18 months and 3 years of age, followed by gradual loss of ambulation, increasing dependence in daily activities, and the development of serious cardiac, respiratory, and orthopedic complications later in life.

In addition to motor impairments, dystrophin deficiency in the brain has been associated with cognitive, behavioral, and psychosocial difficulties. DMD-related mutations affect multiple dystrophin isoforms that are expressed in key brain regions involved in attention, memory, executive functions, and emotional regulation. As a result, children with DMD frequently present with impairments in attention, executive functioning, learning, behavior, and emotional regulation. These non-motor manifestations further complicate disease management and have a substantial impact on participation in daily life and overall quality of life for both children and their families.

During disease progression, increasing motor limitations significantly restrict children's engagement in physical activity and increase the likelihood of adopting a sedentary lifestyle. Reduced physical activity contributes to secondary complications related to disuse, such as decreased cardiorespiratory fitness, reduced bone mineral density, increased fatigue, and further functional decline. Therefore, maintaining and supporting physical activity is considered a critical component of comprehensive care in children with DMD. However, the development of effective and sustainable physical activity-related interventions requires a thorough understanding of the factors influencing physical activity behavior in this population.

In typically developing children, physical activity levels are known to be influenced by a wide range of motor and non-motor factors, including physical function, cognitive status, sleep habits, behavioral characteristics, and family-related environmental and psychosocial factors. Although similar interactions are likely to exist in children with DMD, current evidence regarding the multidimensional determinants of physical activity in this population remains limited. In particular, the combined influence of body functions, activity limitations, participation restrictions, and family-related factors has not been sufficiently investigated within a comprehensive conceptual framework.

The International Classification of Functioning, Disability and Health - Children and Youth Version (ICF-CY), developed by the World Health Organization, provides a biopsychosocial model that enables a holistic evaluation of health by considering body functions and structures, activity, participation, and contextual factors. Using the ICF-CY framework allows for the systematic examination of the dynamic interactions between individual and environmental factors that shape physical activity behavior in children with chronic health conditions.

Therefore, the primary aim of this study is to identify the factors affecting physical activity levels in children with Duchenne Muscular Dystrophy within the ICF-CY framework. Specifically, the study will evaluate the influence of posture, functional capacity, ambulatory status, balance, fatigue, gait, and other musculoskeletal parameters, as well as cognitive status, sleep habits and sleep quality, fear of falling, behavioral characteristics, and motivation on children's physical activity levels. In addition, family-related factors-including caregiver sleep quality, parenting style, perceptions of physical activity, stress level, attitudes and perceptions toward daily life events, and perceived disease impact-will be examined to determine their contribution to physical activity behavior.

By adopting a comprehensive ICF-CY-based approach, this study aims to clarify the relative contribution and magnitude of individual, environmental, and psychosocial factors influencing physical activity levels in children with DMD. The findings are expected to provide clinically relevant insights that may guide the development of targeted, family-centered, and multidimensional interventions aimed at maintaining or enhancing physical activity and improving long-term health outcomes and quality of life in children with Duchenne Muscular Dystrophy.

ELIGIBILITY:
* Inclusion Criteria (Parents):

  1. Being a parent or primary caregiver of a child diagnosed with Duchenne Muscular Dystrophy (DMD),
  2. Volunteering to participate in the study.
* Exclusion Criteria (Parents):

  1. Having caregiving responsibilities for another child or adult with a disability, other than the child with DMD,
  2. Experiencing difficulties in understanding or responding to the questionnaires administered by the physiotherapist.
* Inclusion Criteria (Children with DMD):

  1. Having a confirmed diagnosis of Duchenne Muscular Dystrophy (DMD),
  2. Being between 6 and 14 years of age,
  3. Being classified within the first four levels of the Brooke Lower Extremity Functional Classification (ambulatory children),
  4. Scoring >24 on the Modified Mini-Mental State Examination,
  5. Volunteering to participate in the study.
* Exclusion Criteria (Children with DMD):

  1. Having undergone any musculoskeletal surgery or sustained an injury that could affect physical activity within the past 6 months,
  2. Experiencing difficulty in understanding the test instructions administered by the physiotherapist and therefore being unable to appropriately perform the tests (performance-based assessments),
  3. Experiencing difficulties in understanding or responding to the questionnaires administered by the physiotherapist.

Ages: 6 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Individuals of all self-identified genders are eligible to participate in the study.
Study Population: The study population will consist of children diagnosed with Duchenne Muscular Dystrophy (DMD) and their parents or primary caregivers. Eligible children will be males aged 6 to 14 years with a confirmed diagnosis of DMD who are ambulatory, classified within the first four levels of the Brooke Lower Extremity Functional Classification, and able to follow assessment instructions. Parents or primary caregivers of these children who voluntarily agree to participate will also be included. Participants will be recruited from pediatric neuromuscular rehabilitation and physiotherapy settings.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Children-PAQ-C | At baseline (single assessment at enrollment)
  The physical activity level of children with DMD will be assessed using the Physical Activity Questionnaire for Children (PAQ-C).
The New York Posture Rating Chart | At baseline (single assessment at enrollment)
  The New York Posture Rating Chart will be used to assess posture in children with DMD.
Six Minute Walk Test (6MWT) | At baseline (single assessment at enrollment)
  The 6MWT will be used to evaluate functional capacity in children with DMD.
Pediatric Quality of Life Inventory - Multidimensional Fatigue Scale (PedsQL-MFS) | At baseline (single assessment at enrollment)
  Fatigue in children with DMD will be assessed using the PedsQL-MFS.
Duchenne Muscular Dystrophy Gait Assessment Scale (DMD-GAS) | At baseline (single assessment at enrollment)
  Gait characteristics of children with DMD will be evaluated using the DMD-GAS.
North Star Ambulatory Assessment (NSAA) | At baseline (single assessment at enrollment)
  Ambulatory status of children with DMD will be assessed using the NSAA.
Four Square Step Test (FSST) | At baseline (single assessment at enrollment)
  Balance in children with DMD will be evaluated using the FSST.
Lower Extremity Muscle Strength Assessment | At baseline (single assessment at enrollment)
  Myometric measurements will be performed to assess lower extremity muscle strength in children with DMD.
Assessment of Lower Extremity Joint Range of Motion | At baseline (single assessment at enrollment)
  Active and passive range of motion of the lower extremity joints will be assessed using goniometric measurements.
Muscle Shortness Assessment | At baseline (single assessment at enrollment)
  Muscle length tests will be applied to determine muscle shortness in children with DMD.
Modified Mini-Mental State Examination (MMSE) | At baseline (single assessment at enrollment)
  The Modified MMSE will be used to determine the cognitive level of children with DMD.
Trail Making Test | At baseline (single assessment at enrollment)
  The Trail Making Test will be used to assess cognitive functions such as attention, planning, and executive functions in children with DMD.
Children's Sleep Habits Questionnaire (CSHQ) - Short Form | At baseline (single assessment at enrollment)
  The CSHQ will be used to assess sleep problems in children with DMD.
Pediatric Sleep Questionnaire - Sleep-Related Breathing Disorder Subscale (PSQ-SRBD) | At baseline (single assessment at enrollment)
  The PSQ-SRBD subscale will be used to evaluate sleep-related breathing disorders in children with DMD.
ICF-Based Fear of Falling Form for Pediatric Neuromuscular Diseases (Ped-FOF) | At baseline (single assessment at enrollment)
  The Ped-FOF will be used to assess fear of falling in children with DMD.
Strengths and Difficulties Questionnaire (SDQ) | At baseline (single assessment at enrollment)
  Behavioral problems in children with DMD will be assessed using the SDQ.
Pediatric Motivation Scale (PMS) | At baseline (single assessment at enrollment)
  Motivation levels of children with DMD will be assessed using the PMS.
Pittsburgh Sleep Quality Index (PSQI) | At baseline (single assessment at enrollment)
  Parental sleep quality will be evaluated using the PSQI.
Parenting Scale | At baseline (single assessment at enrollment)
  The Parenting Scale will be used to assess parents' disciplinary practices.
Perceived Barriers to Physical Activity Scale | At baseline (single assessment at enrollment)
  Parents' perceived barriers to participation in physical activity will be assessed using the Perceived Barriers to Physical Activity Scale.
Perceived Stress Scale (PSS) | At baseline (single assessment at enrollment)
  Parental stress levels will be assessed using the PSS.
Cognitive Control and Flexibility Scale (CCFS) | At baseline (single assessment at enrollment)
  The CCFS will be used to assess parents' cognitive flexibility in stressful situations.
Impact on Family Scale (IPFAM) | At baseline (single assessment at enrollment)
  The level of disease-related impact on parents will be assessed using the IPFAM.